CLINICAL TRIAL: NCT05831774
Title: Intraosseous vs. Intravenous Vancomycin Administration in Total Shoulder Arthroplasty: Changing the Paradigm
Brief Title: IO Vancomycin in TSA
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The Methodist Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Patrick McCulloch,MD, Principal Investigator, The Methodist Hospital Research Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRO00036529
Record Dates: First submitted 2023-03-10; First posted 2023-04-26 (Actual); Results first posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Shoulder Injuries
Keywords: total shoulder arthroplasty
MeSH Terms: conditions — Shoulder Injuries | interventions — Jupiter

STUDY DESIGN:
Intervention Model Description: 2 groups - one control, one treatment
Who Masked: Participant, Investigator
Masking Description: Double blinded study
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control - Standard IV administration of vancomycin (Placebo Comparator): Patients will receive the Houston Methodist Hospital orthopedic surgeon's standard of care pre-operative antibiotic regimen for primary total shoulder arthroplasty patients. This includes IV abx (typically ancef or cefepime and vancomycin) will be started in the pre-operative period approximately 1 hour prior to incision (vancomycin dose weight-based at approximately 15mg/kg [6,7] generally 1000-1750mg in 500mL NS).
  Interventions: Drug: Control - Standard IV administration of vancomycin
- Intervention - Intraosseous (IO) administration of vancomycin (Experimental): * IV antibiotics (per physician's standard of care): Typically ancef or cefepime is started in pre-op within 1 hour of incision
  * IO vancomycin is administered in the OR after sterile prep and draping has occurred (500mg in 100-150mL NS).
  * Injection will take place into the proximal humerus
  Interventions: Drug: Intervention - Intraosseous (IO) administration of vancomycin

INTERVENTIONS:
Drug: Intervention - Intraosseous (IO) administration of vancomycin — * IV antibiotics (per physician's standard of care): Typically ancef or cefepime is started in pre-op within 1 hour of incision
  * IO vancomycin is administered in the OR after sterile prep and draping has occurred (500mg in 100-150mL NS).
  * Injection will take place into the proximal humerus
  Arms: Intervention - Intraosseous (IO) administration of vancomycin
Drug: Control - Standard IV administration of vancomycin — Patients will receive the Houston Methodist Hospital orthopedic surgeon's standard of care pre-operative antibiotic regimen for primary total shoulder arthroplasty patients. This includes IV abx (typically ancef or cefepime and vancomycin) will be started in the pre-operative period approximately 1 hour prior to incision (vancomycin dose weight-based at approximately 15mg/kg [6,7] generally 1000-1750mg in 500mL NS).
  Arms: Control - Standard IV administration of vancomycin

SUMMARY:
The purpose of this study is to compare two different antibiotic regimens and techniques during total shoulder arthroplasty.

Primary Objective: Comparable levels of vancomycin will be found in bone, soft tissue, and systemic samples between patient groups.

Secondary Objective: Compare 30 day and 90 day post-operative complication rates (infection) between the control (standard IV administration of vancomycin) vs the interventional group (intraosseous administration of vancomycin). The investigators hypothesize that there will be no difference in complication (infection) rates between groups.

DETAILED DESCRIPTION:
This study is a prospective, randomized, single-blinded, controlled trial. 20 patients in each treatment arm: 20 patients will be given IV vancomycin, 20 patients will be given IO vancomycin. This sample size is based on previous studies examining vancomycin concentration in tourniquetless primary total knee arthroplasty between IO vs IV [12,13].

Once the participant has been enrolled, they will be randomized into either the control group or the experimental group by an excel-based software program prior to their procedure.

Control - Standard IV administration of vancomycin

1) Patients will receive the Houston Methodist Hospital orthopedic surgeon's standard of care pre-operative antibiotic regimen for primary total shoulder arthroplasty patients. This includes IV abx (typically ancef or cefepime and vancomycin) will be started in the pre-operative period approximately 1 hour prior to incision (vancomycin dose weight-based at approximately 15mg/kg [6,7] generally 1000-1750mg in 500mL NS).

Intervention - Intraosseous (IO) administration of vancomycin

1. IV antibiotics (per physician's standard of care): Typically ancef or cefepime is started in pre-op within 1 hour of incision
2. IO vancomycin is administered in the OR after sterile prep and draping has occurred (500mg in 100-150mL NS).
3. Injection will take place into the proximal humerus

All patients in both groups will be monitored during the surgery and immediately post-operatively for adverse injection reactions (i.e. Red Man Syndrome) as this is the standard of care.

All patients (IV and IO) will otherwise follow identical post-operative protocols (including post-operative antibiotic administration)

Intra-Op Sample Collection

Samples will be taken from the following locations at the following times:

Systemic Sample - Start of Case A vancomycin blood level will be drawn by the anesthesiologist staff (CRNA, MD) at the start of incision and should occur simultaneously with the final soft tissue sample collection below Soft tissue sample - Synovium Start A small soft tissue sample will be taken from the synovium upon entering the shoulder joint. This sample will only be taken if it is readily available for the surgeon to gather.

Bone Sample - Bone from Humeral Head After the humeral neck is cut with the "cookie cutter" instrument a portion of humeral head/neck will be removed and placed in a separate specimen jar (remainder of head will be sent to pathology as usual).

Soft Tissue Sample - Synovium End A small soft tissue sample will be taken from the synovium prior to initiation of wound closure. This sample will only be taken if it is readily available for the surgeon to gather.

Systemic Sample A vancomycin blood level will be drawn by the anesthesiologist staff (CRNA, MD) at the time of initiation of closure and should occur simultaneously with the final soft tissue sample collection above

Data Variables to be Recorded Age (calculated from DOB), date of surgery, discharge date, sex, laterality, study group, pre-op creatinine, post-op creatinine, systemic vancomycin level at incision, soft tissue vancomycin level (synovium start and synovium end), humeral head bone sample vancomycin level, and systemic vancomycin level at initiation of wound closure. Additionally, adverse local/systemic reactions as determined from patient's chart, 30-day complications, 90-day complications, cost, time from antibiotic administration to incision, operative time, and incision time.

ELIGIBILITY:
Inclusion Criteria

* Patient is undergoing anatomic or reverse shoulder arthroplasty
* Patient is able to give informed consent to participate on the study. LAR consents will not be utilized for this study
* Age Range >18

Exclusion Criteria:

* Previous shoulder surgery
* BMI above 35
* Contraindication to receiving vancomycin, cefepime, ancef, or other standard of care pre-operative antibiotic (allergy, medical issue, etc).
* Inability to administer the IO infusion
* Refusal to participate
* Diabetes
* Immunocompromised or immunosuppressed patients (HIV, Hep C, ESRD, dialysis, transplant, chemo/radiation treatment in last 6 months, medications)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2026-03-10 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Houston Methodist Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
We do not plan to share this information.

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention - Intraosseous (IO) Administration of Vancomycin: * IV antibiotics (per physician's standard of care): Typically ancef or cefepime is started in pre-op within 1 hour of incision
  * IO vancomycin is administered in the OR after sterile prep and draping has occurred (500mg in 100-150mL NS).
  * Injection will take place into the proximal humerus
  Intervention - Intraosseous (IO) administration of vancomycin: • IV antibiotics (per physician's standard of care): Typically ancef or cefepime is started in pre-op within 1 hour of incision
  * IO vancomycin is administered in the OR after sterile prep and draping has occurred (500mg in 100-150mL NS).
  * Injection will take place into the proximal humerus
Period: Overall Study
Arm/Group | Control - Standard IV Administration of Vancomycin | Intervention - Intraosseous (IO) Administration of Vancomycin
Started | 18 | 15
Completed | 18 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control - Standard IV Administration of Vancomycin | Intervention - Intraosseous (IO) Administration of Vancomycin | Total
Number analyzed (Participants) | 18 | 15 | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 3 | 9
  >=65 years | 12 | 12 | 24
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 5 | 13
  Male | 10 | 10 | 20
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Systemic Levels of Vancomycin
Description: Comparable levels of vancomycin will be found in systemic samples between patient groups.
Time Frame: 24 hours
Population: Please note that these numbers will differ from the participant flow module because one sample from one of the participants was not usable. There was a processing error with the sample in the lab, so values were not obtained.
Measure: Mean (Standard Error); unit: ug/mL
Arm/Group | Control - Standard IV Administration of Vancomycin | Intervention - Intraosseous (IO) Administration of Vancomycin
Number analyzed (Participants) | 17 | 15
ug/mL | 23.65 (3.85) | 9.79 (0.52)

2. Primary Outcome: Vancomycin Levels in the Initial Deltoid
Description: Comparable levels of vancomycin will be found in the initial deltoid samples between patient groups.
Time Frame: 24 hours
Population: as for outcome 1
Measure: Mean (Standard Error); unit: ug/mL
Arm/Group | Control - Standard IV Administration of Vancomycin | Intervention - Intraosseous (IO) Administration of Vancomycin
Number analyzed (Participants) | 17 | 15
ug/mL | 32.7 (4.48) | 31.09 (3.84)

3. Primary Outcome: Vancomycin Levels in the Humeral Head
Description: Comparable levels of vancomycin will be found in humeral head samples between patient groups.
Time Frame: 24 hours
Population: as for outcome 1
Measure: Mean (Standard Error); unit: ug/mL
Arm/Group | Control - Standard IV Administration of Vancomycin | Intervention - Intraosseous (IO) Administration of Vancomycin
Number analyzed (Participants) | 17 | 15
ug/mL | 69.53 (7.71) | 66.5 (8.18)

4. Primary Outcome: Levels of Vancomycin in Synovium
Description: Comparable levels of vancomycin will be found in synovium samples between patient groups.
Time Frame: 24 hours
Population: as for outcome 1
Measure: Mean (Standard Error); unit: ug/mL
Arm/Group | Control - Standard IV Administration of Vancomycin | Intervention - Intraosseous (IO) Administration of Vancomycin
Number analyzed (Participants) | 17 | 15
ug/mL | 34.96 (5.55) | 31.1 (4.7)

5. Primary Outcome: Levels of Vancomycin in Labrum
Description: Comparable levels of vancomycin will be found in labrum samples between patient groups.
Time Frame: 24 hours
Population: as for outcome 1
Measure: Mean (Standard Error); unit: ug/mL
Arm/Group | Control - Standard IV Administration of Vancomycin | Intervention - Intraosseous (IO) Administration of Vancomycin
Number analyzed (Participants) | 17 | 15
ug/mL | 85 (10.87) | 63.54 (6.84)

6. Primary Outcome: Levels of Vancomycin in Glenoid Reaming
Description: Comparable levels of vancomycin will be found in glenoid reaming samples between patient groups.
Time Frame: 24 hours
Population: as for outcome 1
Measure: Mean (Standard Error); unit: ug/mL
Arm/Group | Control - Standard IV Administration of Vancomycin | Intervention - Intraosseous (IO) Administration of Vancomycin
Number analyzed (Participants) | 17 | 15
ug/mL | 67.97 (9.63) | 68.52 (8.92)

7. Primary Outcome: Levels of Vancomycin in Bicep Tendon
Description: Comparable levels of vancomycin will be found in bicep tendon samples between patient groups.
Time Frame: 24 hours
Population: as for outcome 1
Measure: Mean (Standard Error); unit: ug/mL
Arm/Group | Control - Standard IV Administration of Vancomycin | Intervention - Intraosseous (IO) Administration of Vancomycin
Number analyzed (Participants) | 17 | 15
ug/mL | 95.25 (12.54) | 63 (9.05)

8. Primary Outcome: Levels of Vancomycin in End Deltoid
Description: Comparable levels of vancomycin will be found in end deltoid samples between patient groups.
Time Frame: 24 hours
Population: as for outcome 1
Measure: Mean (Standard Error); unit: ug/mL
Arm/Group | Control - Standard IV Administration of Vancomycin | Intervention - Intraosseous (IO) Administration of Vancomycin
Number analyzed (Participants) | 17 | 15
ug/mL | 43.23 (5.48) | 38.68 (5.47)

9. Primary Outcome: Vancomycin Levels in Bicep Tendon
Description: Comparable levels of vancomycin will be found in bicep tendon samples between patient groups.
Time Frame: 24 hours
Population: as for outcome 1
Measure: Mean (Standard Error); unit: ug/mL
Arm/Group | Control - Standard IV Administration of Vancomycin | Intervention - Intraosseous (IO) Administration of Vancomycin
Number analyzed (Participants) | 17 | 15
ug/mL | 95.25 (12.54) | 63 (9.05)

10. Secondary Outcome: Post-operative Complication (Infection) Rates
Description: Compare 30 day and 90 day post-operative complication rates (infection) between the control (standard IV administration of vancomycin) vs the interventional group (intraosseous administration of vancomycin). The investigators hypothesize that there will be no difference in complication (infection) rates between groups.
Time Frame: 30 days, 90 days
Population: as for outcome 1
Measure: Number; unit: Postoperative Complications
Arm/Group | Control - Standard IV Administration of Vancomycin | Intervention - Intraosseous (IO) Administration of Vancomycin
Number analyzed (Participants) | 17 | 15
Postoperative Complications
  30 Days Post-Op | 1 | 0
  90 Days Post-Op | 0 | 0

ADVERSE EVENTS:
Time Frame: Through 90 days postop
Arm/Group | Control - Standard IV Administration of Vancomycin | Intervention - Intraosseous (IO) Administration of Vancomycin
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/15
Other Adverse Events (participants affected / at risk) | 0/18 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-31): https://cdn.clinicaltrials.gov/large-docs/74/NCT05831774/Prot_SAP_000.pdf